CLINICAL TRIAL: NCT00326560
Title: Comparison of Cut and Paste With Sutured Autograft Pterygium Excision
Brief Title: Comparison of Glue With Sutures for Pterygium Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wellington Hospital (Other Government)
Collaborators: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEN/06/03/021
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-06-16 (Estimated); Status verified 2006-05

CONDITIONS: Pterygium
Keywords: Pterygium excision; Cut and paste; Tisseel fibrin glue; Conjunctival autograft
MeSH Terms: conditions — Pterygium

INTERVENTIONS:
Procedure: Pterygium excision and conjunctival autograft

SUMMARY:
Pterygium excision surgery involves excising the abnormal growth from the cornea and filling the defect with a conjunctival (white of the eye) graft from the superior part of the eye. This is the best method of pterygium excision but it is recognised that in 10-15% of cases it will grow back (recurrence). Currently the investigators use small sutures to sew the graft in place. Recently it has been described that glue can be used instead of the sutures. It has been shown in one study that the patient discomfort is less and so is the surgical time. The investigators want to confirm these findings and also compare the recurrence rate between the two types of surgery. They plan to complete a prospective, randomised, control trial of 40 participants. Twenty will have traditional pterygium surgery with the conjunctival autograft sutured. Twenty will have cut and paste surgery with Tisseel glue. The two groups of participants will be compared for pain and discomfort, surgery time, and recurrence rate of the pterygia.

DETAILED DESCRIPTION:
This is a prospective, randomised, control trial of 40 participants. Twenty patients in each arm. Twenty patients undergo standard pterygium excision with the conjunctival autograft sutured. Twenty patients undergo pterygium surgery with Tisseel glue replacing sutures as a method of attaching the conjunctival autograft. Participants will be reviewed, selected, and consented on a pre-assessment day. Surgery will be performed 10 at a time on an all day surgery operating list. Randomisation of the surgery type will be done at the time of surgery after the pterygium has been excised and the autograft taken. One surgeon (R. Hall) will perform all of the procedures. Follow-up will occur at week 1, 2, 4, 26, 52. A questionnaire answered by participants will indicate their pain, foreign body sensation, tearing, and discomfort. There will be observation of any complications such as graft failure and recurrence rate. Photographs will be taken pre-op and post-op.

ELIGIBILITY:
Inclusion Criteria:

* Primary pterygium

Exclusion Criteria:

* Ocular surface disease
* Previous pterygium surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05; Study Completion 2007-09

PRIMARY OUTCOMES:
Surgery time
Patient discomfort at day one, week one, two, four
Recurrence rate at months three, six, twelve

CONTACTS AND LOCATIONS:
Overall Officials: Reece C Hall, MBChB, Principal Investigator — Capital Coast District Health Board
Locations (1):
- Wellington Ophthalmology Department, Capital Coast District Health Board, Wellington, New Zealand

REFERENCES:
- [Background] Koranyi G, Seregard S, Kopp ED. The cut-and-paste method for primary pterygium surgery: long-term follow-up. Acta Ophthalmol Scand. 2005 Jun;83(3):298-301. doi: 10.1111/j.1600-0420.2005.00465.x. PMID 15948780
- [Background] Uy HS, Reyes JM, Flores JD, Lim-Bon-Siong R. Comparison of fibrin glue and sutures for attaching conjunctival autografts after pterygium excision. Ophthalmology. 2005 Apr;112(4):667-71. doi: 10.1016/j.ophtha.2004.08.028. PMID 15808260
- [Background] Koranyi G, Seregard S, Kopp ED. Cut and paste: a no suture, small incision approach to pterygium surgery. Br J Ophthalmol. 2004 Jul;88(7):911-4. doi: 10.1136/bjo.2003.032854. PMID 15205236
- [Derived] Hall RC, Logan AJ, Wells AP. Comparison of fibrin glue with sutures for pterygium excision surgery with conjunctival autografts. Clin Exp Ophthalmol. 2009 Aug;37(6):584-9. doi: 10.1111/j.1442-9071.2009.02105.x. PMID 19702708